CLINICAL TRIAL: NCT07178444
Title: Evaluation of the Effectiveness of an Interdisciplinary Intervention After Acute Coronary Syndrome on Low-Density Lipoprotein Cholesterol Levels
Acronym: EDUSCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP240952; 2025-A00698-41 (Other: French National Agency for the Safety of Medicines and Health Products (ANSM)); PHRIP-23-0025 (Other: French ministry of health, DGOS)
Record Dates: First submitted 2025-08-08; First posted 2025-09-17 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Acute Coronary Syndromes (ACS); Acute Coronary Syndromes
Keywords: acute coronary syndrome; dyslipidemias; patient education; multidisciplinary care team; nurse practitioners
MeSH Terms: conditions — Acute Coronary Syndrome; Dyslipidemias | interventions — Nutritionists; Pharmacists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Standard" care pathway (Active Comparator): Control arm:
  * The French National Health Authority recommends two medical visits (at 6 and 12 month) and, if necessary, a third one (between the first and third month post-ACS) for the monitoring of the left ventricular.
  * The European Society of Cardiology recommends a reassessment of the lipid profile within 4-6 weeks post-ACS.
  Interventions: Other: "Standard" care pathway
- "New" care pathway (Experimental): Intervention arm:
  In addition to the Standard care pathway:
  * One interdisciplinary consultation approximately 4 weeks post-ACS
  * Three consultations with the advanced practice nurse at approximately 3 months, 6 months and 12 months post-ACS
  Interventions: Behavioral: "New" care pathway

INTERVENTIONS:
Behavioral: "New" care pathway — Initially, the patient will have an interdisciplinary consultation aimed at identifying personalized goals for the patient and providing educational/preventive care using tools that will be provided to all centers. This consultation will bring together a cardiologist, an advanced practice nurse (APN), a dietitian and a pharmacist. This consultation will take place approximately 4 weeks after the hospitalization for acute coronary syndrome (ACS).
  Secondly, the patient will have 3 follow-up consultations with the APN (at 3, 6 and 12 months after discharge from hospitalization for an ACS). During these consultations, the APN will perform a clinical assessment, a personalized educational support, a coaching based on the patient's personalized goals, an adjustment of therapies and, depending on needs, referral to other health professionals.
  Other Names: Interdisciplinaire consultation; Identifying personalized goals; Educational/preventive care; Advanced practice nurse; Dietitian; Pharmacist; Acute coronary syndrome; Follow-up consultations with an advanced practice nurse; Coaching; Adjustement of therapies; Coordination of the care pathway
  Arms: "New" care pathway
Other: "Standard" care pathway — The French National Health Authority recommends two medical visits (at 6 and 12 month) and, if necessary, a third one (between the first and third month post-ACS) for the monitoring of the left ventricular. - The European Society of Cardiology recommends a reassessment of the lipid profile within 4-6 weeks post-ACS.
  Arms: "Standard" care pathway

SUMMARY:
According to the World Health Organization (WHO), cardiovascular diseases are the worldwide leading cause of death. For the French public health, cardiovascular diseases are the leading cause of death for the women and the second for men. Each year in France, approximately 120,000 acute coronary syndromes (ACS) occur, including 60,000 myocardial infarctions and more than 15,000 deaths. To prevent or reverse this process, the WHO recommends early detection of the diseases and reduce behavioral and cardiovascular risk factors.

For the patient, the European Society of Cardiology (ESC) recommends the implementation of secondary prevention measures, the lifestyle modifications and the encouragement to become an actor in the management of his health. The first year, the medical follow-up is recommended at 3, 6 and 12 months.

Since 2019, in order to reduce the impact of LDL cholesterol, the ESC has recommended that LDL cholesterol levels be lower than 0.55 g/L accompanied by a reduction of at least 50% from their initial value. In 2023, it clarified this recommendation by recommending a laboratory reassessment within 4-6 weeks after hospital discharge.

The application of these recommendations comes up against the difficulties of real life:

1. The increase in the number of elderly people and people with one or more chronic diseases;
2. In France, the significant regional disparities in the number of physicians;
3. In 2022, six months after hospitalization for an ACS, only 21.6% of French patients had benefited from a cardiac rehabilitation program;
4. Within 12 months of acute coronary syndrome, only 20% to 40% of patients achieved the LDL cholesterol targets recommended by the ESC.

Given the difficulties in implementing the recommendations, investigators believe it is essential to rethink the care pathway for post-ACS patients.

The investigator's hypothesis is that, in addition to the standard pathway, a care offering access to other healthcare professionals (advanced practice nurse, dietitian, pharmacist) should increase the proportion of patients achieving LDL cholesterol targets (LDL cholesterol < 0.55 g/L and a 50% reduction in this level compared to the baseline value) at 12 months. LDL cholesterol was selected as the endpoint because it has been proven that a reduction in LDL cholesterol corresponds to a 22% reduction in cardiovascular events.

To test this hypothesis, the investigators designed a multicenter controlled and randomized trial with two parallel arms:

* "Routine Cares" arm: Each center will program cares as usual and will schedule patient follow-up according to their wishes (cardiac rehabilitation, visits to the general practitioner and/or cardiologist).
* "Intervention" arm: In addition to routine care as described above, the patient will receive an interdisciplinary consultation one month after hospital discharge and three consultations with the IPA (3, 6, and 12 months).

In order for the conclusions of this protocol to reflect French practices, it is planned to include 230 people who have presented with acute coronary syndrome in four healthcare facilities in France (both in Paris and outside Paris).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized for ACS (ST+ or ST-), affiliated with a social security scheme, able to understand the protocol and having signed the study consent.

Exclusion Criteria:

* Patients with a complication of the ACS (mechanical complication, cardiogenic shock, very severe left ventricular dysfunction, presence of an intraventricular thrombus, complex ventricular rhythm disorder) ;
* Proven cognitive impairment or decompensated psychological/psychiatric disorder ;
* Any progressive inflammatory and/or infectious condition ;
* Any orthopedic problem precluding the physical activity ;
* Current participation in any clinical research project aimed at reducing LDL cholesterol levels ;
* Pregnant or breastfeeding woman ;
* Patient receiving state medical assistance ;
* Patient under guardianship or curatorship, or any other legal protection measure ;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reaching the LDL cholesterol target | At enrollment then at the 12th month
  The target is definde as LDL cholesterol level <0.55 g/L and >50% reduction from baseline

SECONDARY OUTCOMES:
Proportion of patients reaching the LDL cholesterol target | At enrollment then at the first month, 6th month and 12th month
  The target for this outcome is defined as LDL cholesterol <0.55 g/L
Proportion of patients reaching the LDL cholesterol target | At enrollment then at the first month, 6th month and 12th month
  The target for this outcome is defined as LDL cholesterol level reduction > 50% compared to baseline value
Changes in cardiovascular risk factors | At enrollment then at the first month, 6th month and 12th month
  This outcome aims to assess changes in the patient's overall cardiovascular risk profile throughout the study. Multiple parameters will be evaluated to capture a comprehensive picture of the modifications in cardiovascular risk factors presented by each patient. The parametrers will be:
  * Dyslipidemia: Proportion of patients achieving the LDL cholesterol target set by the European Society of Cardiology (<0.55 g/L and >50% reduction from baseline)
  * Hypertension: Proportion of patients achieving a systolic blood pressure < 140 mmHg and a diastolic blood pressure < 90 mmHg
  * Percentage of patients with controlled type 2 diabetes (for a diabetic patient, HbA1c target <7%)
  * BMI
Physical Activity Score | At enrollment then at the 6th month and 12th month
  Total score on the "Ricci and Gagnon Self-Assessment of Physical Activity" Questionnaire (activity self-assessment questionnaire).
  The minimum value is 9 The maximum value is 45 Under 18: inactive Between 18 and 35: active Over 35: very active
Proportion of patients who participated in a cardiac rehabilitation program | At 6th month and 12th month
  This outcome aims to assess the proportion of patients who engage in a cardiac rehabilitation program following an acute coronary syndrome
Proportion of patients consuming toxic substances and their quantity measured | At enrollment then at the 6th month and 12th month
  The substances involved are: alcohol, tobacco, and drugs
Quality of life score | At enrollment then at the 6th month and 12th month
  Measured using the EQ-5D-5L Questionnaire (European quality of life 5 dimensions 5 levels questionnaire) The (EQ-5D-5L) questionnaire provides two types of scores. The first is an index scored derived from five health dimensions (mobility, self-care, actual activities, pain/discomfort, and anxiety/depression) converted into a single value ranged from 0 (representing health states considered worse than death) to 1(representing perfect health). The second is the EQ Visual Analogue Scale (EQ-VAS), a self-rated health measure ranging from 0 ("the worst health you can imagine") to 100 ("the best health you can imagine") representing self-rated health.
Therapeutic Compliance Score | At enrollment then at the 6th month and 12th month
  Measured using FREEDOM questionnaire (FREE Detection non Observance Medication) The FREEDOM questionnaire includes 11 items rated on a 4-point Likert scale ranging from "strongly disagree" to "strongly agree". The questionnaire responses will be used qualitatively, without calculation of a numerical total score, to classify patients into categories of medication adherence (low, moderate, high).
List of lipid-lowering treatments taken by patients | At enrollment then at the first month, 6th month and 12th month
  This outcome aims to describe the lipid-lowering therapy prescribed to each patient, as well as any modifications made during follow-up. This outcome focuses solely on documenting which lipid-lowering treatments patients are receiving and does not involve any comparison or evaluation of the effectiveness or safety of different lipid-lowering therapie
Number of medical (cardiologist or general practitioner) and/or paramedical (dietician, etc.) consultations | At 6th month and 12th month
Mortality rate and the reasons | At 6th month and 12th month
Rehospitalization rates and the reasons | At 6th month and 12th month
Rate of cardiovascular events | At 12th month
Estimation of cost per QALY gained and cost per serious cardiac event avoided | At 12th month
  QALY: quality-adjusted life year
Professional satisfaction rate by using a satisfaction scale from 0 to 10 | At 12th month
  Satisfaction with the care provided to the patient under the EDUSCA protocol

CONTACTS AND LOCATIONS:
Overall Officials: Melissa JOLY GOURJAULT, Principal Investigator — Hôpital Européen Georges Pompidou - AP-HP; Thibaut CARUBA, Study Chair — Hôpital européen Georges-Pompidou - AP-HP
Locations (4):
- France (4):
  - Centre Hospitalier Sud Francilien, Pôle Cardiologie, Corbeil-Essonnes
  - Hopital Saint Joseph-Saint Luc, Cardiologie, Lyon
  - CHU Montpellier - Hôpital Arnaud de Villeneuve, Cardiologie, Montpellier
  - Hôpital Européen Georges Pompidou - AP-HP, Cardiologie, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).